CLINICAL TRIAL: NCT07390071
Title: Multimodal Telerehabilitation in Patients Undergoing CAR-T Cell Immunotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HCI190212
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma; Myeloma; Cytokine Release Syndrome; Immune Effector Cell Associated Neurotoxicity Syndrome
MeSH Terms: conditions — Lymphoma; Neoplasms, Plasma Cell; Cytokine Release Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multimodal Cancer Telerehabilitation (Experimental): Each enrolled patient will undergo a four-week multimodal prehabilitation before the commencement of the CAR-T therapy. During CAR-T therapy, the patients will use an interactive app supporting cancer self-care education and early mobilization while undergoing chemotherapy, infusion, in-hospital toxicity monitoring, and recovery (the duration depends on the specific CAR-T treatment regimen). After completion of the CAR-T procedures and hospital discharge, the patients will undergo a 12-week home-based multimodal telerehabilitation.
  Individualized rehabilitation plans using a web-based care management portal. Patients at home follow a safe and effective personalized exercise and nutrition plan guided by interactive touch-screen technology combined with behavioral counseling, social support, and interactive education and empowerment.
  Interventions: Device: Home Automated Telemanagement (HAT) Patient Unit

INTERVENTIONS:
Device: Home Automated Telemanagement (HAT) Patient Unit — HAT (Home Automated Telemanagement) patient unit will guide patients in following their treatment plans, including exercise and diet prescriptions, monitor patients' progress and symptoms, and communication with health care providers.
  Participants will receive an internet-enabled device, either a touchscreen tablet or a virtual reality (VR) headset, as part of the patient unit, based on their personal preference. Participants will also be provided a pulse oximeter to monitor their heart rate and oxygen saturation, and a fitbit to assess daily physical activity and step counts.

SUMMARY:
The proposed multimodal telerehabilitation model allows a rehabilitation therapy team to set up individualized rehabilitation plans using a web-based care management portal and monitor patient progress online. Patients at home follow a safe and effective personalized exercise and nutrition plan guided by interactive touch-screen technology combined with behavioral counseling, social support, and interactive education and empowerment. The design of the telerehabilitation system is based on the cloud-based Internet-of-Things architecture allowing real-time monitoring of cardiovascular parameters and exercise performance. The patient's level of exertion during exercise is automatically identified by a validated AI-driven algorithm supporting exercise safety and efficacy. The ultimate goal of this pilot feasibility project is to establish the extent of the impact of the proposed patient-centered cancer telerehabilitation model on disease-specific quality of life, and functional and symptom outcomes and to obtain sufficient evidence for a definitive randomized clinical trial evaluating this approach in a multi-center study.

DETAILED DESCRIPTION:
CAR-T therapy is a relatively new, innovative treatment strategy to manage refractory hematological cancers, including some types of leukemia, lymphoma, and multiple myeloma (Efficace, 2022). This pivotal treatment has become a standard-of-care for certain malignancies, such as relapsed non-Hodgkins lymphoma, relapsed or refractory acute lymphoblastic leukemia, and relapsed refractory multiple myeloma, with some studies showing at least 80% of the patients with a positive response to treatment (June, 2018; Landry, 2020). While CAR T-cell therapy has led to significant advances in the treatment of hematologic malignancies, it also presents a set of unique toxicities. The two most common acute adverse effects are cytokine release syndrome (CRS) and neurological toxicity known as immune effector cell-associated neurotoxicity syndrome (ICANS), respectively (Neelapu, 2017).

Recent studies suggest that there should be an emphasis on prehabilitation soon after initiating the workup process for CAR-T therapy, maintaining function during active treatment, and close follow-up with rehabilitation especially if neurological sequelae persist (Obaisi, 2022; Kiefer, 2023). Effective interventions are urgently needed to improve the QoL and functional capacity in patients with hematological cancers undergoing CAR-T therapy (Cenik, 2020;Jeevanantham, 2021). Physical activity programs have been shown to impact psychological symptoms, fatigue, and quality of life (Vermaete, 2013, 2014). Crucially, no evidence has been presented to date for patients with hematologic malignancies while undergoing CAR-T therapy. Thus, studies exploring approaches to expand access to multimodal cancer rehabilitation practices in these patients are necessary to address the needs of the rapidly growing population of cancer survivors receiving CAR-T therapy. Recent systematic reviews demonstrated the high potential of telehealth approaches to facilitate cancer rehabilitation (Brick, 2022; Chang, 2022).

Home Automated Telemanagement (HAT). The HAT system is a telemedicine platform supporting patients in following individualized self-care plans and assisting healthcare practitioners in the treatment and monitoring of their patients according to evidence-based guidelines (Finkelstein, 2012; Fleg, 2020; Shero, 2022). HAT is based on the chronic disease care model (Grover, 2014) and provides support for patient self-management, comprehensive patient-provider communication, and multidisciplinary care coordination (Drouin, 2015). The main objective of the HAT system is to minimize the burden of chronic disease management and to simplify monitoring in ambulatory care. To achieve this goal, the HAT system is required (1) to support a constant information feedback loop between the patient and health care providers; (2) to take over all routine repetitive tasks; and (3) to provide real-time clinical decision support both for the patient and clinician. HAT has been successfully implemented and tested in a variety of chronic diseases.

Patient units are used at patient homes to guide patients in following their treatment plans including exercise and diet prescriptions, monitor patients' progress and symptoms, and to communicate with health care providers. Any web-enabled device can serve as a patient unit including touchscreen tablets, VR headsets, and smartphones. The home unit interface underwent rigorous usability testing (Jeong, 2015; Finkelstein, 2021; Gabriel, 2023) and is very simple to operate, even by those without any prior computer experience. The clinician units (any web-enabled device) are used to set up and update individualized treatment plans, analyze patient self-testing results, and review computer-generated alerts. The HAT server implements computerized decision support based on individualized alert setup and realtime monitoring of patient self-testing data. In this study, the HAT system will be focused on the delivery of a multimodal cancer rehabilitation program comprising individualized therapeutic physical exercise, nutrition plan, behavioral counseling, and tailored educational empowerment targeting the social, cognitive, reproductive, and vocational needs of blood cancer survivors.

The proposed multimodal telerehabilitation model allows a rehabilitation therapy team to set up individualized rehabilitation plans using a web-based care management portal and monitor patient progress online. Patients at home follow a safe and effective personalized exercise and nutrition plan guided by interactive touch-screen technology combined with behavioral counseling, social support, and interactive education and empowerment. The design of the telerehabilitation system is based on the cloud-based Internet-of-Things architecture allowing real-time monitoring of cardiovascular parameters and exercise performance. The patient's level of exertion during exercise is automatically identified by a validated AI-driven algorithm supporting exercise safety and efficacy. The ultimate goal of this pilot feasibility project is to establish the extent of the impact of the proposed patient-centered cancer telerehabilitation model on disease-specific quality of life, and functional and symptom outcomes and to obtain sufficient evidence for a definitive randomized clinical trial evaluating this approach in a multi-center study.

This study will determine if patients with hematologic malignancies undergoing CAR-T therapy will demonstrate sufficient acceptability and adherence to the multimodal cancer telerehabilitation, and it will be associated with a positive trajectory of QoL, fitness, and patient-reported outcomes. This trial is an exploratory sequential mixed methods design to assess the feasibility of a patient-centered, culturally tailored telemedicine approach for multimodal cancer rehabilitation in patients with hematologic malignancies undergoing CAR-T therapy.

Eligible patients will undergo a four-week multimodal prehabilitation before the commencement of the CAR-T therapy and then receive continuous online empowerment and education support during CAR-T therapy while undergoing chemotherapy, CAR-T infusion, toxicity monitoring, and recovery for up to four weeks, depending on a specific CAR-T treatment regimen. This will be followed by a twelve-week multimodal telerehabilitation after treatment completion and hospital discharge. A comprehensive assessment will be conducted at the beginning of the study, and the patients will be individually prescribed resistance, aerobic, and relaxation exercises, and a nutrition plan for 4-week prehabilitation based on patient fitness levels and nutrition status. A mobile app will provide interactive education on cancer survivorship, early mobilization, and post-discharge self-care during CAR-T treatment comprising outpatient chemotherapy, CART infusion, and in-patient hospitalization for toxicity monitoring. After the hospital discharge, a 12-week multimodal rehabilitation plan will be provided via the telerehabilitation system which uses validated AI-driven real-time assessment of exercise exertion (Smiley, 2024). Social support will be delivered via group telecounseling sessions. Automated analysis of daily exercise and nutrition logs will alert the telerehabilitation team about low patient adherence and prompt tailored feedback by the telerehabilitation team. The acceptability, usability, feasibility, and adherence will be assessed at the end of the study as described in the Analysis Plan. Finally, this study will assess QoL, fitness, body composition, cancer symptoms, behavioral characteristics, and satisfaction with care before and after the multimodal rehabilitation delivered via a telemedicine platform.

ELIGIBILITY:
Inclusion Criteria:

* age >21
* confirmed diagnosis of lymphoma or myeloma
* commercial FDA-approved CAR-T delivery planned for ≥4 weeks following enrollment
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Access to a working telephone line in their home or a cell phone.

Exclusion Criteria:

* have unstable angina, uncontrolled hypertension, recent myocardial infarction, pacemakers, painful or unstable bony metastases, or recent skeletal fractures;
* are engaged in a regular exercise rehabilitation program;
* have relocation plans within next 6 months;
* participate in another clinical trial.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
System Usability Score - Feasibility | up to 12 weeks after completion of the CAR-T procedures.
  To assess the feasibility of a multimodal cancer telerehabilitation model in patients with hematologic malignancies undergoing CAR-T therapy by evaluating system usability, acceptability, and exercise adherence. This outcome measure will report the System Usability Score for home telerehabilitation in patients undergoing CAR-T therapy.
  The System Usability Scale (SUS) is a 10-item, 5-point Likert questionnaire that yields a single usability score on a 0-100 scale; the minimum possible score is 0 (worst perceived usability) and the maximum is 100 (best perceived usability). This outcome measure will report the mean System Usability Score at 12 weeks after completion of the CAR-T procedure.
Adherence Indicators - Feasibility | up to 12 weeks after completion of the CAR-T procedures.
  To assess the feasibility of a multimodal cancer telerehabilitation model in patients with hematologic malignancies undergoing CAR-T therapy by evaluating daily exercise logs. This outcome measure will report adherence based on daily exercise logs in patients utilizing the home telerehabilitation after undergoing CAR-T therapy.
  Adherence will be defined as the percentage of exercise sessions of the total number of prescribed exercise sessions.

SECONDARY OUTCOMES:
6-minute walk distance (6MWD) | up to 12 weeks after completion of the CAR-T procedures.
  6MWD is an assessment of functional and aerobic capacity by measuring how far a patient can walk over 6 minutes.
  This outcome measure will report mean 6MWD.
Short Physical Performance Battery (SPPB) | up to 12 weeks after completion of the CAR-T procedures.
  The Short Physical Performance Battery (SPPB) is a series of assessments to measure balance, strength, and physical functioning. SPPB scores range from 0-12, with lower scores indicating severe limitations and higher scores indicating better physical functioning.
  This outcome measure will report mean SPPB.
Godin Leisure Score Index | up to 12 weeks after completion of the CAR-T procedures.
  Godin Leisure Score Index is a questionnaire to assess time spent in leisure exercise. Godin Leisure Score Index is a continuous index, with a minimum of 0. Lower scores indicate lower activity and higher cores indicate higher activity.
  This outcome measure will report mean Godin Leisure Score Index.
Extended Activities of Daily Living (ADL) | up to 12 weeks after completion of the CAR-T procedures.
  The Extended ADL scale is an assessment of functional independence. Extended ADL is a 22-item questionnaire, with each item scaled from 0 to 3.
  The Extended ADL total score ranges from 0 to 66, with lower scores indicating better functional independence and higher scores indicating worse functional independence.
36-Item Short Form Survey (SF-36) | up to 12 weeks after completion of the CAR-T procedures.
  SF-36 is a questionnaire that assesses patient health. This outcome measure will report 8 sub-scores: physical function, pain, limitations due to physical health issues, limitations due to personal/emotional issues, emotional well-being, social functioning, energy/fatigue, and general health perceptions.
  Each sub-score ranges from 0-100, with higher score indicating more favorable health and lower score indicating less favorable health.
European Organization For Research And Treatment Of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | up to 12 weeks after completion of the CAR-T procedures.
  EORTC QLQ-C30 is a questionnaire to assess health-related quality of life in cancer patients. Patients indicate which symptoms/problems they have experienced during the past week, from "1 Not at All" to "4 Very Much".
  The assessment will report data as 15 subscales with scores from 0-100. A high score indicates a higher response level.
  A high functional scale score (FS) represents a high/healthy level of function and includes Physical, Role, Emotional, Cognitive, and Social functioning. A high symptom scale score (SS) represent a high level of symptomatology/problems and includes Fatigue, Nausea and vomiting, Pain, Dyspnoea, Insomnia, Appetite loss, Constipation, Diarrhoea, Financial difficulties, and Global health status/QoL.
  This outcome will report the mean score of each subscale.
Functional Assessment of Cancer Therapy-Fatigue (FACT-F) | up to 12 weeks after completion of the CAR-T procedures.
  The FACT-F is a self-reported evaluation of fatigue in cancer patients. This questionnaire has patients rank statements regarding Physical, Social/Family, Emotional, and Functional well-being and Fatigue from 0 "Not at All" to 4 "Very Much".
  The FACT-F has a minimum of 0 and a maximum of 52, with higher scores indicating less fatigue and lower scores indicating more fatigue.
Numeric Rating Scale (NRS) | up to 12 weeks after completion of the CAR-T procedures.
  NRS is a single-item question assessing pain. NRS scores range from 0-10, with lower scores indicating less pain and higher scores indicating more pain.
  This outcome measure will report mean NRS.
Exercise Self-Efficacy Scale (EXSE) | up to 12 weeks after completion of the CAR-T procedures.
  The EXSE assesses exercise self-efficacy, or a patient's belief in their ability to continue regular exercise.
  Outcome Expectations for Exercise Scale is an 8-item questionnaire. Each item is a 10-point scale, ranging from 0% (NOT AT ALL CONFIDENT) to 100% (Highly CONFIDENT).
  Total score ranges from 0 to 100, with lower scores indicating worse exercise self-efficacy and higher scores indicating better exercise self-efficacy.
Behavioral Regulation in Exercise Questionnaire 3 (BREQ-3) | up to 12 weeks after completion of the CAR-T procedures.
  BREQ-3 is an assessment measuring a patient's exercise motivation. BREQ-3 reports 6 sub-scores: Amotivation and External, Introjected, Identified, Integrated, and Intrinsic regulation.
  BREQ-3 score ranges from 0 to 96. Lower scores indicate lower motivation, and higher scores indicate higher motivation.
  This outcome measure will report the mean BREQ-3.
Outcome Expectations for Exercise Scale | up to 12 weeks after completion of the CAR-T procedures.
  The Outcome Expectations for Exercise Scale assesses beliefs and attitudes about the benefits of exercise.
  Outcome Expectations for Exercise Scale is a 15-item questionnaire. Each item is a 5-point Likert scale, ranging from 1 (strongly disagree) to 5 (strongly agree).
  Total score ranges from 15 to 75, with lower scores indicating worse exercise attitudes and higher scores indicating better exercise attitudes.
Medical Outcome Study (MOS) Exercise Adherence Questionnaire | up to 12 weeks after completion of the CAR-T procedures.
  The MOS Exercise Adherence Questionnaire assesses patient adherence to exercise.
  MOS Exercise Adherence Questionnaire is a 40-item questionnaire. Scores range from 0 to 100, with lower scores indicating worse exercise adherence and higher scores indicating better exercise adherence.
Telerehab user attitudes | up to 12 weeks after completion of the CAR-T procedures.
  Telerehab user attitudes measure patients' overall feelings about remote rehabilitation technology and service. The minimum possible score is 11 (worst perceived attitude) and the maximum is 55 (best perceived attitude).
  This outcome measure will report the mean Telerehab user attitudes at 12 weeks after completion of the CAR-T procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Sborov, MD, MS, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Acharya UH, Dhawale T, Yun S, Jacobson CA, Chavez JC, Ramos JD, Appelbaum J, Maloney DG. Management of cytokine release syndrome and neurotoxicity in chimeric antigen receptor (CAR) T cell therapy. Expert Rev Hematol. 2019 Mar;12(3):195-205. doi: 10.1080/17474086.2019.1585238. Epub 2019 Mar 18. PMID 30793644
- [Background] Alfano CM, Cheville AL, Mustian K. Developing High-Quality Cancer Rehabilitation Programs: A Timely Need. Am Soc Clin Oncol Educ Book. 2016;35:241-9. doi: 10.1200/EDBK_156164. PMID 27249704
- [Background] AlJohi AA, Aljehani GH, AlSaeed SA, Alhoqail H, Mohammed J, Madi SM. Evidence-based exercises intervention in adults diagnosed with Lymphoma. Saudi Med J. 2022 May;43(5):441-450. doi: 10.15537/smj.2022.43.5.20210894. PMID 35537731
- [Background] Amatya B, Khan F, Lew TE, Dickinson M. Rehabilitation in patients with lymphoma: An overview of Systematic Reviews. J Rehabil Med. 2021 Mar 17;53(3):jrm00163. doi: 10.2340/16501977-2810. PMID 33710351
- [Background] Amireault S, Godin G, Lacombe J, Sabiston CM. The use of the Godin-Shephard Leisure-Time Physical Activity Questionnaire in oncology research: a systematic review. BMC Med Res Methodol. 2015 Aug 12;15:60. doi: 10.1186/s12874-015-0045-7. PMID 26264621
- [Background] Barnett-Page E, Thomas J. Methods for the synthesis of qualitative research: a critical review. BMC Med Res Methodol. 2009 Aug 11;9:59. doi: 10.1186/1471-2288-9-59. PMID 19671152
- [Background] Bedra M, Wick E, Brotman D, Finkelstein J. Avatar-based interactive ileostomy education in hospitalized patients. Stud Health Technol Inform. 2013;190:83-5. PMID 23823383
- [Background] Bedra M, McNabney M, Stiassny D, Nicholas J, Finkelstein J. Defining patient-centered characteristics of a telerehabilitation system for patients with COPD. Stud Health Technol Inform. 2013;190:24-6. PMID 23823363
- [Background] Bedra M, Finkelstein J. Feasibility of post-acute hip fracture telerehabilitation in older adults. Stud Health Technol Inform. 2015;210:469-73. PMID 25991191
- [Background] Benzo R. Satori: Awakening to Outcomes That Matter: The Impact of Social Support in Chronic Obstructive Pulmonary Disease. Ann Am Thorac Soc. 2017 Sep;14(9):1385-1386. doi: 10.1513/AnnalsATS.201707-526ED. No abstract available. PMID 28862500
- [Background] Blanchard CM, Courneya KS, Rodgers WM, Murnaghan DM. Determinants of exercise intention and behavior in survivors of breast and prostate cancer: an application of the theory of planned behavior. Cancer Nurs. 2002 Apr;25(2):88-95. doi: 10.1097/00002820-200204000-00002. PMID 11984095
- [Background] Borrell-Vega J, Esparza Gutierrez AG, Humeidan ML. Multimodal Prehabilitation Programs for Older Surgical Patients. Anesthesiol Clin. 2019 Sep;37(3):437-452. doi: 10.1016/j.anclin.2019.04.004. Epub 2019 Jun 26. PMID 31337477
- [Background] Brennan L, Sheill G, O'Neill L, O'Connor L, Smyth E, Guinan E. Physical Therapists in Oncology Settings: Experiences in Delivering Cancer Rehabilitation Services, Barriers to Care, and Service Development Needs. Phys Ther. 2022 Mar 1;102(3):pzab287. doi: 10.1093/ptj/pzab287. PMID 35084029
- [Background] Brick R, Padgett L, Jones J, Wood KC, Pergolotti M, Marshall TF, Campbell G, Eilers R, Keshavarzi S, Flores AM, Silver JK, Virani A, Livinski AA, Ahmed MF, Kendig T, Khalid B, Barnett J, Borhani A, Bernard G, Lyons KD. The influence of telehealth-based cancer rehabilitation interventions on disability: a systematic review. J Cancer Surviv. 2023 Dec;17(6):1725-1750. doi: 10.1007/s11764-022-01181-4. Epub 2022 Feb 26. PMID 35218521
- [Background] Brooke J. SUS: A quick and dirty usability scale. Usability Eval. Ind., 1995:189.
- [Background] Burton M, Valet M, Caty G, Aboubakar F, Reychler G. Telerehabilitation physical exercise for patients with lung cancer through the course of their disease: A systematic review. J Telemed Telecare. 2024 Jun;30(5):756-780. doi: 10.1177/1357633X221094200. Epub 2022 May 12. PMID 35546542
- [Background] Bustoros M, Mouhieddine TH, Detappe A, Ghobrial IM. Established and Novel Prognostic Biomarkers in Multiple Myeloma. Am Soc Clin Oncol Educ Book. 2017;37:548-560. doi: 10.1200/EDBK_175175. PMID 28561668
- [Background] Capelan M, Battisti NML, McLoughlin A, Maidens V, Snuggs N, Slyk P, Peckitt C, Ring A. The prevalence of unmet needs in 625 women living beyond a diagnosis of early breast cancer. Br J Cancer. 2017 Oct 10;117(8):1113-1120. doi: 10.1038/bjc.2017.283. Epub 2017 Aug 31. PMID 28859057
- [Background] Cappell KM, Kochenderfer JN. Long-term outcomes following CAR T cell therapy: what we know so far. Nat Rev Clin Oncol. 2023 Jun;20(6):359-371. doi: 10.1038/s41571-023-00754-1. Epub 2023 Apr 13. PMID 37055515
- [Background] Cenik F, Keilani M, Hasenohrl T, Huber D, Stuhlpfarrer B, Pataraia A, Crevenna R. Relevant parameters for recommendations of physical activity in patients suffering from multiple myeloma : A pilot study. Wien Klin Wochenschr. 2020 Mar;132(5-6):124-131. doi: 10.1007/s00508-019-01582-z. Epub 2019 Nov 29. PMID 31784826
- [Background] Chan ZY, Lim CF, Leow JL, et al. Using the technology acceptance model to examine acceptance of telemedicine by cancer patients in an ambulatory care setting. Proceedings of Singapore Healthcare 2022;31:1-11.
- [Background] Chang P, Zheng J. Updates in Cancer Rehabilitation Telehealth. Curr Phys Med Rehabil Rep. 2022;10(4):332-338. doi: 10.1007/s40141-022-00372-5. Epub 2022 Nov 9. PMID 36408472
- [Background] Cheville AL, Kornblith AB, Basford JR. An examination of the causes for the underutilization of rehabilitation services among people with advanced cancer. Am J Phys Med Rehabil. 2011 May;90(5 Suppl 1):S27-37. doi: 10.1097/PHM.0b013e31820be3be. PMID 21765261
- [Background] Cocks K, Wells JR, Johnson C, Schmidt H, Koller M, Oerlemans S, Velikova G, Pinto M, Tomaszewski KA, Aaronson NK, Exall E, Finbow C, Fitzsimmons D, Grant L, Groenvold M, Tolley C, Wheelwright S, Bottomley A; European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Group. Content validity of the EORTC quality of life questionnaire QLQ-C30 for use in cancer. Eur J Cancer. 2023 Jan;178:128-138. doi: 10.1016/j.ejca.2022.10.026. Epub 2022 Nov 1. PMID 36436330
- [Background] Courneya KS, Sellar CM, Stevinson C, McNeely ML, Peddle CJ, Friedenreich CM, Tankel K, Basi S, Chua N, Mazurek A, Reiman T. Randomized controlled trial of the effects of aerobic exercise on physical functioning and quality of life in lymphoma patients. J Clin Oncol. 2009 Sep 20;27(27):4605-12. doi: 10.1200/JCO.2008.20.0634. Epub 2009 Aug 17. PMID 19687337
- [Background] Cross RK, Cheevers N, Rustgi A, Langenberg P, Finkelstein J. Randomized, controlled trial of home telemanagement in patients with ulcerative colitis (UC HAT). Inflamm Bowel Dis. 2012 Jun;18(6):1018-25. doi: 10.1002/ibd.21795. Epub 2011 Jun 17. PMID 21688350
- [Background] Damschroder LJ, Lowery JC. Evaluation of a large-scale weight management program using the consolidated framework for implementation research (CFIR). Implement Sci. 2013 May 10;8:51. doi: 10.1186/1748-5908-8-51. PMID 23663819
- [Background] Damschroder LJ, Reardon CM, Widerquist MAO, Lowery J. The updated Consolidated Framework for Implementation Research based on user feedback. Implement Sci. 2022 Oct 29;17(1):75. doi: 10.1186/s13012-022-01245-0. PMID 36309746
- [Background] Damschroder LJ, Reardon CM, Opra Widerquist MA, Lowery J. Conceptualizing outcomes for use with the Consolidated Framework for Implementation Research (CFIR): the CFIR Outcomes Addendum. Implement Sci. 2022 Jan 22;17(1):7. doi: 10.1186/s13012-021-01181-5. PMID 35065675
- [Background] das Nair R, Moreton BJ, Lincoln NB. Rasch analysis of the Nottingham extended activities of daily living scale. J Rehabil Med. 2011 Oct;43(10):944-50. doi: 10.2340/16501977-0858. PMID 21879232
- [Background] de Fatima Ribeiro Silva C, Ohara DG, Matos AP, Pinto ACPN, Pegorari MS. Short Physical Performance Battery as a Measure of Physical Performance and Mortality Predictor in Older Adults: A Comprehensive Literature Review. Int J Environ Res Public Health. 2021 Oct 10;18(20):10612. doi: 10.3390/ijerph182010612. PMID 34682359
- [Background] Drouin H, Walker J, McNeil H, Elliott J, Stolee P. Measured outcomes of chronic care programs for older adults: a systematic review. BMC Geriatr. 2015 Oct 26;15:139. doi: 10.1186/s12877-015-0136-7. PMID 26503159
- [Background] Duque E, Fonseca G, Vieira H, Gontijo G, Ishitani L. A systematic literature review on user centered design and participatory design with older people. IHC '19: Proceedings of the 18th Brazilian Symposium on Human Factors in Computing Systems, October 2019, Article No. 9, pp. 1-11, doi.org/10.1145/3357155.3358471.
- [Background] Eaves YD. A synthesis technique for grounded theory data analysis. J Adv Nurs. 2001 Sep;35(5):654-63. doi: 10.1046/j.1365-2648.2001.01897.x. PMID 11529967
- [Background] Edward J, Petermann VM, Eberth JM, Zahnd WE, Vanderpool RC, Askelson N, Rohweder CL, Gonzalez SK, Stradtman LR, Ko LK, Farris PE. Interventions to address cancer-related financial toxicity: Recommendations from the field. J Rural Health. 2022 Sep;38(4):817-826. doi: 10.1111/jrh.12637. Epub 2021 Dec 3. PMID 34861066
- [Background] Efficace F, Cannella L, Sparano F, Giesinger JM, Vignetti M, Baron F, Bruera E, Luppi M, Platzbecker U. Chimeric Antigen Receptor T-cell Therapy in Hematologic Malignancies and Patient-reported Outcomes: A Scoping Review. Hemasphere. 2022 Dec 1;6(12):e802. doi: 10.1097/HS9.0000000000000802. eCollection 2022 Dec. PMID 36504547
- [Background] Elliott J, Fallows A, Staetsky L, Smith PW, Foster CL, Maher EJ, Corner J. The health and well-being of cancer survivors in the UK: findings from a population-based survey. Br J Cancer. 2011 Nov 8;105 Suppl 1(Suppl 1):S11-20. doi: 10.1038/bjc.2011.418. PMID 22048028
- [Background] Faithfull S, Turner L, Poole K, Joy M, Manders R, Weprin J, Winters-Stone K, Saxton J. Prehabilitation for adults diagnosed with cancer: A systematic review of long-term physical function, nutrition and patient-reported outcomes. Eur J Cancer Care (Engl). 2019 Jul;28(4):e13023. doi: 10.1111/ecc.13023. Epub 2019 Mar 11. PMID 30859650
- [Background] Finkelstein J, Cabrera MR, Hripcsak G. Internet-based home asthma telemonitoring: can patients handle the technology? Chest. 2000 Jan;117(1):148-55. doi: 10.1378/chest.117.1.148. PMID 10631213
- [Background] Finkelstein J, Amelung P. Quality of Life in Asthma Patients is Affected by Home Telemanagement. Value in Health 2005;8(3):246.
- [Background] Finkelstein J, Lapshin O. Reducing depression stigma using a web-based program. Int J Med Inform. 2007 Oct;76(10):726-34. doi: 10.1016/j.ijmedinf.2006.07.004. Epub 2006 Sep 20. PMID 16996299
- [Background] Finkelstein J, Lapshin O, Wasserman E. Randomized study of different anti-stigma media. Patient Educ Couns. 2008 May;71(2):204-14. doi: 10.1016/j.pec.2008.01.002. Epub 2008 Mar 4. PMID 18289823
- [Background] Finkelstein J, Lapshin O, Castro H, Cha E, Provance PG. Home-based physical telerehabilitation in patients with multiple sclerosis: a pilot study. J Rehabil Res Dev. 2008;45(9):1361-73. PMID 19319760
- [Background] Finkelstein J, Lapshin O, Cha E. Feasibility of promoting smoking cessation among methadone users using multimedia computer-assisted education. J Med Internet Res. 2008 Nov 3;10(5):e33. doi: 10.2196/jmir.1089. PMID 18984556
- [Background] Finkelstein J, Cha E. Hypertension telemanagement in blacks. Circ Cardiovasc Qual Outcomes. 2009 May;2(3):272-8. doi: 10.1161/CIRCOUTCOMES.109.849968. PMID 20031848
- [Background] Finkelstein J, Wood J, Cha E, Orlov A, Dennison C. Feasibility of congestive heart failure telemanagement using a wii-based telecare platform. Annu Int Conf IEEE Eng Med Biol Soc. 2010;2010:2211-4. doi: 10.1109/IEMBS.2010.5627087. PMID 21096432
- [Background] Finkelstein J, Wood J. Information technology for continuous patient health education. Proceedings of the 2011 Conference on Information Technology Education (SIGITE '11), 2011, pp. 245-250, doi: 10.1145/2047594.2047658.
- [Background] Finkelstein J, Wood J. Universal Platform for Individualized Continuous Patient Education (iCOPE). Proceedings of the IASTED International Conference on Technology for Education (TE 2011), 2011, pp. 24-30, doi: 10.2316/P.2011.754-025.
- [Background] Finkelstein J, Wood J. Using individualized continuous patient education (iCOPE) platform to facilitate smoking cessation in hospitalized patients. 2012 International Symposium on Information Technologies in Medicine and Education, Hokkaido, Japan, 2012, pp. 727-731, doi: 10.1109/ITiME.2012.6291406.
- [Background] Finkelstein J, Wood J, Cha E. Impact of physical telerehabilitation on functional outcomes in seniors with mobility limitations. Annu Int Conf IEEE Eng Med Biol Soc. 2012;2012:5827-32. doi: 10.1109/EMBC.2012.6347319. PMID 23367254
- [Background] Finkelstein J, Cha E, Wood J, Wallin MT. Predictors of successful acceptance of home telemanagement in veterans with Multiple Sclerosis. Annu Int Conf IEEE Eng Med Biol Soc. 2013;2013:7314-7. doi: 10.1109/EMBC.2013.6611247. PMID 24111434
- [Background] Finkelstein J, Jeong Ic. Remotely controlled cycling exercise system for home-based telerehabilitation. Annu Int Conf IEEE Eng Med Biol Soc. 2013;2013:7310-3. doi: 10.1109/EMBC.2013.6611246. PMID 24111433
- [Background] Finkelstein J, Jeong IC. Design and Implementation of Home Automated Telemanagement Platform for Interactive Biking Exercise (iBikE HAT). Proc. of the IEEE-EMBS Special Topic Conference on Point-of-Care Healthcare Technologies (POCHT2013), 2013, pp. 236-239.
- [Background] Finkelstein J, Cha E, Royal W. Predictors of Acceptance of Using Games for Cognitive Rehabilitation. Int J of MS Care 2013;15(Suppl 3):35.
- [Background] Finkelstein J, Bedra M. Is Internet search better than structured instruction for web-based health education? Stud Health Technol Inform. 2013;190:65-7. PMID 23823377
- [Background] Finkelstein J, Jeong IC. Feasibility of interactive biking exercise system for telemanagement in elderly. Stud Health Technol Inform. 2013;192:642-6. PMID 23920635
- [Background] Finkelstein J, Cisse P, Jeong IC. Feasibility of Interactive Resistance Chair in Older Adults with Diabetes. Stud Health Technol Inform. 2015;213:61-4. PMID 26152953
- [Background] Finkelstein J, Bedra M. Avatar-based Interactive Diabetes Education in Older Adults. Journal of the American Geriatrics Society 2015;62:S64.
- [Background] Finkelstein J, Bedra M, Li X, Wood J, Ouyang P. Mobile App to Reduce Inactivity in Sedentary Overweight Women. Stud Health Technol Inform. 2015;216:89-92. PMID 26262016
- [Background] Finkelstein J, Cha EM. Using a Mobile App to Promote Smoking Cessation in Hospitalized Patients. JMIR Mhealth Uhealth. 2016 May 6;4(2):e59. doi: 10.2196/mhealth.5149. PMID 27154792
- [Background] Finkelstein J, Wood J, Crew KD, Kukafka R. Introducing a Comprehensive Informatics Framework to Promote Breast Cancer Risk Assessment and Chemoprevention in the Primary Care Setting. AMIA Jt Summits Transl Sci Proc. 2017 Jul 26;2017:58-67. eCollection 2017. PMID 28815107
- [Background] Finkelstein J, Doerstling M, Rocco P, Karpatkin H. Remote exercise capacity assessment in home-based telerehabilitation. Archives of Physical Medicine and Rehabilitation 2021;102(4):e4-e5.
- [Background] Finkelstein J, Huo X, Parvanova I, Galsky M. Usability Inspection of a Mobile Cancer Telerehabilitation System. Stud Health Technol Inform. 2022 Jan 14;289:405-409. doi: 10.3233/SHTI210944. PMID 35062177
- [Background] Finkelstein J, Parvanova I, Huo X. Feasibility of a Virtual Reality App to Promote Pulmonary Rehabilitation. Stud Health Technol Inform. 2023 May 18;302:458-462. doi: 10.3233/SHTI230172. PMID 37203716
- [Background] Finkelstein J, Rocco P. Comprehensive Health Informatics Engagement Framework for Pulmonary Rehabilitation. Archives of Physical Medicine and Rehabilitation 2024;105(4):e138.
- [Background] Fleg JL, Keteyian SJ, Peterson PN, Benzo R, Finkelstein J, Forman DE, Gaalema DE, Cooper LS, Punturieri A, Joseph L, Shero S, Zieman S. Increasing Use of Cardiac and Pulmonary Rehabilitation in Traditional and Community Settings: OPPORTUNITIES TO REDUCE HEALTH CARE DISPARITIES. J Cardiopulm Rehabil Prev. 2020 Nov;40(6):350-355. doi: 10.1097/HCR.0000000000000527. PMID 33074849
- [Background] Gabriel AS, Tsai TY, Xhakli T, Finkelstein J. Mixed-Methods Assessment of a Virtual Reality-Based System for Pulmonary Rehabilitation. Stud Health Technol Inform. 2023 Oct 20;309:245-249. doi: 10.3233/SHTI230789. PMID 37869851
- [Background] Gabriel AS, Parvanova I, Tsai TY, Finkelstein J. Assessing Patient Perspectives of a Cancer Telerehabilitation Platform Using Thematic Analysis of Semi-Structured Qualitative Interviews. AMIA Jt Summits Transl Sci Proc. 2023 Jun 16;2023:216-224. eCollection 2023. PMID 37350908
- [Background] Gabriel AS, Parvanova I, Finkelstein J. Patient Perspectives on Long-Term Use of a Pulmonary Telerehabilitation Platform: A Qualitative Analysis. Stud Health Technol Inform. 2023 May 18;302:982-986. doi: 10.3233/SHTI230322. PMID 37203549
- [Background] Gabriel AS, Tsai TY, Xhakli T, Finkelstein J. Patient Perceptions of a Virtual Reality-Based System for Pulmonary Rehabilitation: A Qualitative Analysis. Stud Health Technol Inform. 2023 Jun 29;305:406-409. doi: 10.3233/SHTI230517. PMID 37387051
- [Background] Gerteis M, Edgman-Levitan S, Daley J, Delbanco TL Through the Patient's Eyes: Understanding and Promoting Patient-Centered Care. San Francisco, CA: Jossey-Bass; 1993.
- [Background] Granger CL. Physiotherapy management of blood cancers. J Physiother. 2023 Apr;69(2):70-78. doi: 10.1016/j.jphys.2023.02.015. Epub 2023 Mar 21. No abstract available. PMID 36958978
- [Background] Graves KD. Social cognitive theory and cancer patients' quality of life: a meta-analysis of psychosocial intervention components. Health Psychol. 2003 Mar;22(2):210-9. PMID 12683741
- [Background] Grimshaw C, Keteyian SJ, Benzo R, Finkelstein J, Forman DE, Gaalema DE, Peterson PN, Einhorn PT, Punturieri A, Shero S, Fleg JL. Baseline Characteristics and Barriers to Recruitment in Cardiac and Pulmonary Rehabilitation NIH-Funded Trials. J Cardiopulm Rehabil Prev. 2023 Nov 1;43(6):407-411. doi: 10.1097/HCR.0000000000000824. Epub 2023 Aug 29. No abstract available. PMID 37643249
- [Background] Grover A, Joshi A. An overview of chronic disease models: a systematic literature review. Glob J Health Sci. 2014 Oct 29;7(2):210-27. doi: 10.5539/gjhs.v7n2p210. PMID 25716407
- [Background] Guo Y, Ding L, Miao X, Jiang X, Xu T, Xu X, Zhu S, Xu Q, Hu J. Effects of prehabilitation on postoperative outcomes in frail cancer patients undergoing elective surgery: a systematic review and meta-analysis. Support Care Cancer. 2022 Dec 19;31(1):57. doi: 10.1007/s00520-022-07541-1. PMID 36534300
- [Background] Hertzog MA. Considerations in determining sample size for pilot studies. Res Nurs Health. 2008 Apr;31(2):180-91. doi: 10.1002/nur.20247. PMID 18183564
- [Background] Holden RJ, Karsh BT. The technology acceptance model: its past and its future in health care. J Biomed Inform. 2010 Feb;43(1):159-72. doi: 10.1016/j.jbi.2009.07.002. Epub 2009 Jul 15. PMID 19615467
- [Background] Holden CE, Wheelwright S, Harle A, Wagland R. The role of health literacy in cancer care: A mixed studies systematic review. PLoS One. 2021 Nov 12;16(11):e0259815. doi: 10.1371/journal.pone.0259815. eCollection 2021. PMID 34767562
- [Background] Holm LV, Hansen DG, Johansen C, Vedsted P, Larsen PV, Kragstrup J, Sondergaard J. Participation in cancer rehabilitation and unmet needs: a population-based cohort study. Support Care Cancer. 2012 Nov;20(11):2913-24. doi: 10.1007/s00520-012-1420-0. Epub 2012 Mar 14. PMID 22415608
- [Background] Hoogland AI, Jayani RV, Collier A, Irizarry-Arroyo N, Rodriguez Y, Jain MD, Booth-Jones M, Hyland KA, James BW, Barata A, Bachmeier CA, Chavez JC, Khimani F, Krivenko GS, Lazaryan A, Liu HD, Nishihori T, Pinilla-Ibarz J, Shah BD, Abidi M, Locke FL, Jim HSL. Acute patient-reported outcomes in B-cell malignancies treated with axicabtagene ciloleucel. Cancer Med. 2021 Mar;10(6):1936-1943. doi: 10.1002/cam4.3664. Epub 2021 Feb 28. PMID 33641257
- [Background] Jeevanantham D, Rajendran V, McGillis Z, Tremblay L, Lariviere C, Knight A. Mobilization and Exercise Intervention for Patients With Multiple Myeloma: Clinical Practice Guidelines Endorsed by the Canadian Physiotherapy Association. Phys Ther. 2021 Jan 4;101(1):pzaa180. doi: 10.1093/ptj/pzaa180. PMID 32975563
- [Background] Jeong Ic, Finkelstein J. Potential value of electrocardiogram and photoplethysmogram for non-invasive blood pressure estimation during exercise. Annu Int Conf IEEE Eng Med Biol Soc. 2013;2013:2304-7. doi: 10.1109/EMBC.2013.6609998. PMID 24110185
- [Background] Jeong IC, Finkelstein J. Classification of cycling exercise status using short-term heart rate variability. Annu Int Conf IEEE Eng Med Biol Soc. 2014;2014:1782-5. doi: 10.1109/EMBC.2014.6943954. PMID 25570322
- [Background] Jeong IC, Finkelstein J. Remotely controlled biking is associated with improved adherence to prescribed cycling speed. Technol Health Care. 2015;23 Suppl 2:S543-9. doi: 10.3233/THC-150992. PMID 26410522
- [Background] Jeong IC, Finkelstein J. Real-Time Classification of Exercise Exertion Levels Using Discriminant Analysis of HRV Data. Stud Health Technol Inform. 2015;213:171-4. PMID 26152984
- [Background] Jeong IC, Finkelstein J. Introducing Contactless Blood Pressure Assessment Using a High Speed Video Camera. J Med Syst. 2016 Apr;40(4):77. doi: 10.1007/s10916-016-0439-z. Epub 2016 Jan 20. PMID 26791993
- [Background] Jeong IC, Karpatkin H, Finkelstein J. Physical Telerehabilitation Improves Quality of Life in Patients with Multiple Sclerosis. Stud Health Technol Inform. 2021 Dec 15;284:384-388. doi: 10.3233/SHTI210752. PMID 34920553
- [Background] Jones JM, Olson K, Catton P, Catton CN, Fleshner NE, Krzyzanowska MK, McCready DR, Wong RK, Jiang H, Howell D. Cancer-related fatigue and associated disability in post-treatment cancer survivors. J Cancer Surviv. 2016 Feb;10(1):51-61. doi: 10.1007/s11764-015-0450-2. Epub 2015 Apr 16. PMID 25876557
- [Background] Joyce DD, Wallis CJD, Huang LC, Hoffman KE, Zhao Z, Koyama T, Goodman M, Hamilton AS, Wu XC, Paddock LE, Stroup A, Cooperberg MR, Hashibe M, O'Neil BB, Kaplan SH, Greenfield S, Penson DF, Barocas DA. The Association Between Financial Toxicity and Treatment Regret in Men With Localized Prostate Cancer. JNCI Cancer Spectr. 2022 Nov 1;6(6):pkac071. doi: 10.1093/jncics/pkac071. PMID 36255249
- [Background] June CH, Sadelain M. Chimeric Antigen Receptor Therapy. N Engl J Med. 2018 Jul 5;379(1):64-73. doi: 10.1056/NEJMra1706169. No abstract available. PMID 29972754
- [Background] Kamal M, Joseph J, Greenbaum U, Hicklen R, Kebriaei P, Srour SA, Wang XS. Patient-Reported Outcomes for Cancer Patients with Hematological Malignancies Undergoing Chimeric Antigen Receptor T Cell Therapy: A Systematic Review. Transplant Cell Ther. 2021 May;27(5):390.e1-390.e7. doi: 10.1016/j.jtct.2021.01.003. Epub 2021 Jan 7. PMID 33965176
- [Background] Kamal SA, Shafiq M, Kakria P. Investigating acceptance of telemedicine services through an extended technology acceptance model (TAM). Technology in Society 2020;60:101212.
- [Background] Kammin EJ. The 6-Minute Walk Test: Indications and Guidelines for Use in Outpatient Practices. J Nurse Pract. 2022 Jun;18(6):608-610. doi: 10.1016/j.nurpra.2022.04.013. Epub 2022 May 12. PMID 35578650
- [Background] Keilani M, Kainberger F, Pataraia A, Hasenohrl T, Wagner B, Palma S, Cenik F, Crevenna R. Typical aspects in the rehabilitation of cancer patients suffering from metastatic bone disease or multiple myeloma. Wien Klin Wochenschr. 2019 Nov;131(21-22):567-575. doi: 10.1007/s00508-019-1524-3. Epub 2019 Jul 2. PMID 31267163
- [Background] Khajouei R, Zahiri Esfahani M, Jahani Y. Comparison of heuristic and cognitive walkthrough usability evaluation methods for evaluating health information systems. J Am Med Inform Assoc. 2017 Apr 1;24(e1):e55-e60. doi: 10.1093/jamia/ocw100. PMID 27497799
- [Background] Kiefer T, Luders C, Voller H, Daeschlein G. Rehabilitation of patients after CAR T-cell therapy. Experiences on 5 patients. Transpl Immunol. 2023 Feb;76:101770. doi: 10.1016/j.trim.2022.101770. Epub 2022 Dec 5. PMID 36470571
- [Background] Kirk MA, Kelley C, Yankey N, Birken SA, Abadie B, Damschroder L. A systematic review of the use of the Consolidated Framework for Implementation Research. Implement Sci. 2016 May 17;11:72. doi: 10.1186/s13012-016-0437-z. PMID 27189233
- [Background] Knips L, Bergenthal N, Streckmann F, Monsef I, Elter T, Skoetz N. Aerobic physical exercise for adult patients with haematological malignancies. Cochrane Database Syst Rev. 2019 Jan 31;1(1):CD009075. doi: 10.1002/14651858.CD009075.pub3. PMID 30702150
- [Background] Lahteenmaki Taalas T, Jarvela L, Niinikoski H, Huurre A, Harila-Saari A. Inflammatory biomarkers after an exercise intervention in childhood acute lymphoblastic leukemia survivors. EJHaem. 2022 Sep 29;3(4):1188-1200. doi: 10.1002/jha2.588. eCollection 2022 Nov. PMID 36467791
- [Background] Lecat CSY, McCourt O, Land J, Yong K, Fisher A. Multiple myeloma and physical activity. BMC Res Notes. 2021 May 7;14(1):171. doi: 10.1186/s13104-021-05591-y. PMID 33962674
- [Background] Lee DW, Gardner R, Porter DL, Louis CU, Ahmed N, Jensen M, Grupp SA, Mackall CL. Current concepts in the diagnosis and management of cytokine release syndrome. Blood. 2014 Jul 10;124(2):188-95. doi: 10.1182/blood-2014-05-552729. Epub 2014 May 29. PMID 24876563
- [Background] Lentz R, Benson AB 3rd, Kircher S. Financial toxicity in cancer care: Prevalence, causes, consequences, and reduction strategies. J Surg Oncol. 2019 Jul;120(1):85-92. doi: 10.1002/jso.25374. Epub 2019 Jan 16. PMID 30650186
- [Background] Levine RL. Healthy People 2030: A Beacon for Addressing Health Disparities and Health Equity. J Public Health Manag Pract. 2021 Nov-Dec 01;27(Suppl 6):S220-S221. doi: 10.1097/PHH.0000000000001409. No abstract available. PMID 34559739
- [Background] Ligibel JA, Bohlke K, May AM, Clinton SK, Demark-Wahnefried W, Gilchrist SC, Irwin ML, Late M, Mansfield S, Marshall TF, Meyerhardt JA, Thomson CA, Wood WA, Alfano CM. Exercise, Diet, and Weight Management During Cancer Treatment: ASCO Guideline. J Clin Oncol. 2022 Aug 1;40(22):2491-2507. doi: 10.1200/JCO.22.00687. Epub 2022 May 16. PMID 35576506
- [Background] Lins L, Carvalho FM. SF-36 total score as a single measure of health-related quality of life: Scoping review. SAGE Open Med. 2016 Oct 4;4:2050312116671725. doi: 10.1177/2050312116671725. eCollection 2016. PMID 27757230
- [Background] Lopez-Bueno R, Andersen LL, Koyanagi A, Nunez-Cortes R, Calatayud J, Casana J, Del Pozo Cruz B. Thresholds of handgrip strength for all-cause, cancer, and cardiovascular mortality: A systematic review with dose-response meta-analysis. Ageing Res Rev. 2022 Dec;82:101778. doi: 10.1016/j.arr.2022.101778. Epub 2022 Nov 1. PMID 36332759
- [Background] McDermott LA, Murphy MH, McNeilly AM, Rankin JP, Gracey JH. Biological markers as an outcome measure of exercise in cancer rehabilitation: A systematic review. J Cancer Res Ther. 2018 Jan-Mar;14(2):267-277. doi: 10.4103/0973-1482.191036. PMID 29516906
- [Background] Meneses-Echavez JF, Loaiza-Betancur AF, Diaz-Lopez V, Echavarria-Rodriguez AM, Triana-Reina HR. Prehabilitation programs for individuals with cancer: a systematic review of randomized-controlled trials. Syst Rev. 2023 Nov 17;12(1):219. doi: 10.1186/s13643-023-02373-4. PMID 37978411
- [Background] Michael CM, Lehrer EJ, Schmitz KH, Zaorsky NG. Prehabilitation exercise therapy for cancer: A systematic review and meta-analysis. Cancer Med. 2021 Jul;10(13):4195-4205. doi: 10.1002/cam4.4021. Epub 2021 Jun 10. PMID 34110101
- [Background] Minns Lowe CJ, Wilson MS, Sackley CM, Barker KL. Blind outcome assessment: the development and use of procedures to maintain and describe blinding in a pragmatic physiotherapy rehabilitation trial. Clin Rehabil. 2011 Mar;25(3):264-74. doi: 10.1177/0269215510380824. Epub 2010 Oct 22. PMID 20971749
- [Background] Nadal C, Sas C, Doherty G. Technology Acceptance in Mobile Health: Scoping Review of Definitions, Models, and Measurement. J Med Internet Res. 2020 Jul 6;22(7):e17256. doi: 10.2196/17256. PMID 32628122
- [Background] Nakano J, Hashizume K, Fukushima T, Ueno K, Matsuura E, Ikio Y, Ishii S, Morishita S, Tanaka K, Kusuba Y. Effects of Aerobic and Resistance Exercises on Physical Symptoms in Cancer Patients: A Meta-analysis. Integr Cancer Ther. 2018 Dec;17(4):1048-1058. doi: 10.1177/1534735418807555. Epub 2018 Oct 23. PMID 30352523
- [Background] Neelapu SS, Locke FL, Bartlett NL, Lekakis LJ, Miklos DB, Jacobson CA, Braunschweig I, Oluwole OO, Siddiqi T, Lin Y, Timmerman JM, Stiff PJ, Friedberg JW, Flinn IW, Goy A, Hill BT, Smith MR, Deol A, Farooq U, McSweeney P, Munoz J, Avivi I, Castro JE, Westin JR, Chavez JC, Ghobadi A, Komanduri KV, Levy R, Jacobsen ED, Witzig TE, Reagan P, Bot A, Rossi J, Navale L, Jiang Y, Aycock J, Elias M, Chang D, Wiezorek J, Go WY. Axicabtagene Ciloleucel CAR T-Cell Therapy in Refractory Large B-Cell Lymphoma. N Engl J Med. 2017 Dec 28;377(26):2531-2544. doi: 10.1056/NEJMoa1707447. Epub 2017 Dec 10. PMID 29226797
- [Background] Nielsen J, Molich R. Heuristic Evaluation of User Interfaces. CHI'90 Proceedings, ACM, 1990, pp. 249-256.
- [Background] Nielsen J. Usability Engineering. Morgan Kaufmann; 1st edition (September 23, 1993). 384 pp.
- [Background] Nielsen J, Mack RL (editors). Usability Inspection Methods; Wiley; 1st edition (May 9, 1994). 448 pp.
- [Background] Obaisi O, Fontillas RC, Patel K, Ngo-Huang A. Rehabilitation Needs for Patients Undergoing CAR T-Cell Therapy. Curr Oncol Rep. 2022 Jun;24(6):741-749. doi: 10.1007/s11912-022-01240-0. Epub 2022 Mar 10. PMID 35267151
- [Background] Oberoi S, Robinson PD, Cataudella D, Culos-Reed SN, Davis H, Duong N, Gibson F, Gotte M, Hinds P, Nijhof SL, Tomlinson D, van der Torre P, Cabral S, Dupuis LL, Sung L. Physical activity reduces fatigue in patients with cancer and hematopoietic stem cell transplant recipients: A systematic review and meta-analysis of randomized trials. Crit Rev Oncol Hematol. 2018 Feb;122:52-59. doi: 10.1016/j.critrevonc.2017.12.011. Epub 2017 Dec 16. PMID 29458789
- [Background] Oechsle K, Aslan Z, Suesse Y, Jensen W, Bokemeyer C, de Wit M. Multimodal exercise training during myeloablative chemotherapy: a prospective randomized pilot trial. Support Care Cancer. 2014 Jan;22(1):63-9. doi: 10.1007/s00520-013-1927-z. Epub 2013 Aug 29. PMID 23989498
- [Background] Oerlemans S, Mols F, Nijziel MR, Lybeert M, van de Poll-Franse LV. The impact of treatment, socio-demographic and clinical characteristics on health-related quality of life among Hodgkin's and non-Hodgkin's lymphoma survivors: a systematic review. Ann Hematol. 2011 Sep;90(9):993-1004. doi: 10.1007/s00277-011-1274-4. Epub 2011 Jun 14. PMID 21670973
- [Background] Oerlemans S, Issa DE, van den Broek EC, Nijziel MR, Coebergh JW, Mols F, van de Poll-Franse LV. Impact of therapy and disease-related symptoms on health-related quality of life in patients with follicular lymphoma: results of the population-based PHAROS-registry. Eur J Haematol. 2014 Sep;93(3):229-38. doi: 10.1111/ejh.12335. Epub 2014 Apr 26. PMID 24702126
- [Background] Oerlemans S, Nijziel MR, van de Poll-Franse LV. Age-related differences in quality of life among patients with diffuse large B-cell lymphoma. Cancer. 2015 Aug 15;121(16):2857-8. doi: 10.1002/cncr.29427. Epub 2015 Apr 29. No abstract available. PMID 25926003
- [Background] Pasek M, Suchocka L, Gasior K. Model of Social Support for Patients Treated for Cancer. Cancers (Basel). 2021 Sep 24;13(19):4786. doi: 10.3390/cancers13194786. PMID 34638270
- [Background] Patel KB, Turner K, Alishahi Tabriz A, Gonzalez BD, Oswald LB, Nguyen OT, Hong YR, Jim HSL, Nichols AC, Wang X, Robinson E, Naso C, Spiess PE. Estimated Indirect Cost Savings of Using Telehealth Among Nonelderly Patients With Cancer. JAMA Netw Open. 2023 Jan 3;6(1):e2250211. doi: 10.1001/jamanetworkopen.2022.50211. PMID 36626174
- [Background] Patrick K, Intille SS, Zabinski MF. An ecological framework for cancer communication: implications for research. J Med Internet Res. 2005 Jul 1;7(3):e23. doi: 10.2196/jmir.7.3.e23. PMID 15998614
- [Background] Pergolotti M, Deal AM, Lavery J, Reeve BB, Muss HB. The prevalence of potentially modifiable functional deficits and the subsequent use of occupational and physical therapy by older adults with cancer. J Geriatr Oncol. 2015 May;6(3):194-201. doi: 10.1016/j.jgo.2015.01.004. Epub 2015 Jan 19. PMID 25614296
- [Background] Persoon S, Kersten MJ, van der Weiden K, Buffart LM, Nollet F, Brug J, Chinapaw MJ. Effects of exercise in patients treated with stem cell transplantation for a hematologic malignancy: a systematic review and meta-analysis. Cancer Treat Rev. 2013 Oct;39(6):682-90. doi: 10.1016/j.ctrv.2013.01.001. Epub 2013 Feb 26. PMID 23485478
- [Background] Priest H, Roberts P, Woods L. An overview of three different approaches to the interpretation of qualitative data. Part 1: Theoretical issues. Nurse Res. 2002;10(1):30-42. doi: 10.7748/nr2002.10.10.1.30.c5877. PMID 12405004
- [Background] Raedeke TD, Dlugonski D. High Versus Low Theoretical Fidelity Pedometer Intervention Using Social-Cognitive Theory on Steps and Self-Efficacy. Res Q Exerc Sport. 2017 Dec;88(4):436-446. doi: 10.1080/02701367.2017.1368976. Epub 2017 Sep 20. PMID 28929950
- [Background] Rangachari P, Mushiana SS, Herbert K. A scoping review of applications of the Consolidated Framework for Implementation Research (CFIR) to telehealth service implementation initiatives. BMC Health Serv Res. 2022 Nov 30;22(1):1450. doi: 10.1186/s12913-022-08871-w. PMID 36447279
- [Background] Ratcliff R, Voskuilen C, McKoon G. Internal and external sources of variability in perceptual decision-making. Psychol Rev. 2018 Jan;125(1):33-46. doi: 10.1037/rev0000080. Epub 2017 Oct 16. PMID 29035076
- [Background] Robins D, Brody R, Jeong IC, Parvanova I, Liu J, Finkelstein J. Towards a Highly Usable, Mobile Electronic Platform for Patient Recruitment and Consent Management. Stud Health Technol Inform. 2020 Jun 16;270:1066-1070. doi: 10.3233/SHTI200325. PMID 32570545
- [Background] Rocco P, Finkelstein J. Telerehabilitation for Patients with Cancer: A Scoping Review. Stud Health Technol Inform. 2022 Jun 6;290:543-546. doi: 10.3233/SHTI220136. PMID 35673075
- [Background] Rubin DB. Multiple imputation after 18+ years (with discussion). Journal of the American Statistical Association 1996;91:473-489.
- [Background] Ruff MW, Siegler EL, Kenderian SS. A Concise Review of Neurologic Complications Associated with Chimeric Antigen Receptor T-cell Immunotherapy. Neurol Clin. 2020 Nov;38(4):953-963. doi: 10.1016/j.ncl.2020.08.001. Epub 2020 Sep 12. PMID 33040871
- [Background] Sacristan JA, Aguaron A, Avendano-Sola C, Garrido P, Carrion J, Gutierrez A, Kroes R, Flores A. Patient involvement in clinical research: why, when, and how. Patient Prefer Adherence. 2016 Apr 27;10:631-40. doi: 10.2147/PPA.S104259. eCollection 2016. PMID 27175063
- [Background] Scheffer DDL, Latini A. Exercise-induced immune system response: Anti-inflammatory status on peripheral and central organs. Biochim Biophys Acta Mol Basis Dis. 2020 Oct 1;1866(10):165823. doi: 10.1016/j.bbadis.2020.165823. Epub 2020 Apr 29. PMID 32360589
- [Background] Schmidt K, Vogt L, Thiel C, Jager E, Banzer W. Validity of the six-minute walk test in cancer patients. Int J Sports Med. 2013 Jul;34(7):631-6. doi: 10.1055/s-0032-1323746. Epub 2013 Feb 26. PMID 23444095
- [Background] Schubert ML, Schmitt M, Wang L, Ramos CA, Jordan K, Muller-Tidow C, Dreger P. Side-effect management of chimeric antigen receptor (CAR) T-cell therapy. Ann Oncol. 2021 Jan;32(1):34-48. doi: 10.1016/j.annonc.2020.10.478. Epub 2020 Oct 21. PMID 33098993
- [Background] Shero ST, Benzo R, Cooper LS, Finkelstein J, Forman DE, Gaalema DE, Joseph L, Keteyian SJ, Peterson PN, Punturieri A, Zieman S, Fleg JL. Update on RFA Increasing Use of Cardiac and Pulmonary Rehabilitation in Traditional and Community Settings NIH-Funded Trials: ADDRESSING CLINICAL TRIAL CHALLENGES PRESENTED BY THE COVID-19 PANDEMIC. J Cardiopulm Rehabil Prev. 2022 Jan 1;42(1):10-14. doi: 10.1097/HCR.0000000000000635. PMID 34508036
- [Background] Shimabukuro-Vornhagen A, Godel P, Subklewe M, Stemmler HJ, Schlosser HA, Schlaak M, Kochanek M, Boll B, von Bergwelt-Baildon MS. Cytokine release syndrome. J Immunother Cancer. 2018 Jun 15;6(1):56. doi: 10.1186/s40425-018-0343-9. PMID 29907163
- [Background] Sidana S, Thanarajasingam G, Griffin J, Thompson CA, Burtis M, Warsame R, et al. Patient experience of chimeric antigen receptor (CAR)-T cell therapy vs. stem cell transplant: longitudinal patient reported adverse events, cognition and quality of life. Blood. 2019;134:794.
- [Background] Siemonsma PC, Walker MF. Practical guidelines for independent assessment in randomized controlled trials (RCTs) of rehabilitation. Clin Rehabil. 1997 Nov;11(4):273-9. doi: 10.1177/026921559701100402. PMID 9408666
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer statistics, 2022. CA Cancer J Clin. 2022 Jan;72(1):7-33. doi: 10.3322/caac.21708. Epub 2022 Jan 12. PMID 35020204
- [Background] Silver JK, Baima J, Mayer RS. Impairment-driven cancer rehabilitation: an essential component of quality care and survivorship. CA Cancer J Clin. 2013 Sep;63(5):295-317. doi: 10.3322/caac.21186. Epub 2013 Jul 15. PMID 23856764
- [Background] Skrabal Ross X, Gunn KM, Olver I. Understanding the strategies rural cancer patients and survivors use to manage financial toxicity and the broader implications on their lives. Support Care Cancer. 2021 Sep;29(9):5487-5496. doi: 10.1007/s00520-021-06086-z. Epub 2021 Mar 12. PMID 33710410
- [Background] Smiley A, Tsai TY, Cui W, Parvanova I, Lyu J, Zakashansky E, Xhakli T, Cui H, Finkelstein J. Telemonitoring of Home-Based Biking Exercise: Assessment of Wireless Interfaces. JMIR Biomed Eng. 2022 Oct 12;7(2):e41782. doi: 10.2196/41782. PMID 38875588
- [Background] Smiley A, Tsai TY, Finkelstein, J. Wireless real-time exercise system for physical telerehabilitation. 2022 IEEE Long Island Systems, Applications, and Technology Conference (LISAT), 2022, pp. 1-6. doi: 10.1109/LISAT50122.2022.9923944.
- [Background] Smiley A, Finkelstein J. Aerobic exercise system for home telerehabilitation. 2022 IEEE 35th International Symposium on Computer-Based Medical Systems (CBMS), 2022, pp. 297-301. doi: 10.1109/CBMS55023.2022.00059.
- [Background] Smiley A, Tsai TY, Zakashansky E, Gabriel A, Xhakli T, Cui W, Huo X, Havrylchuk I, Cui H, Finkelstein J. Exercise Exertion Levels Prediction Based on Real-Time Wearable Physiological Signal Monitoring. Stud Health Technol Inform. 2023 Jun 29;305:172-175. doi: 10.3233/SHTI230454. PMID 37386988
- [Background] Smiley A, Tsai TY, Havrylchuk I, Cui W, Parvanova I, Zakashansky E, Xhakli T, Cui H, Finkelstein J. Development and Evaluation of Wireless Interfaces to Monitor and Control Cycling Exercise During Home Telerehabilitation. Med Devices (Auckl). 2023 Jan 19;16:1-13. doi: 10.2147/MDER.S392999. eCollection 2023. PMID 36698919
- [Background] Smiley A, Finkelstein J. Forecasting Exercise Exertion Levels Using LSTM Modeling of Wearable Physiological Data. 2024 IEEE First International Conference on Artificial Intelligence for Medicine, Health and Care (AIMHC), Laguna Hills, CA, USA, 2024, pp. 173-176, doi: 10.1109/AIMHC59811.2024.00038.
- [Background] Smiley A, Tsai TY, Havrylchuk I, Gabriel A, Zakashansky E, Xhakli T, Lyu J, Cui W, Parvanova I, Finkelstein J. Machine Learning Approaches for Exercise Exertion Level Classification Using Data from Wearable Physiologic Monitors. Stud Health Technol Inform. 2024 Jan 25;310:1428-1429. doi: 10.3233/SHTI231228. PMID 38269680
- [Background] Stacey FG, James EL, Chapman K, Courneya KS, Lubans DR. A systematic review and meta-analysis of social cognitive theory-based physical activity and/or nutrition behavior change interventions for cancer survivors. J Cancer Surviv. 2015 Jun;9(2):305-38. doi: 10.1007/s11764-014-0413-z. Epub 2014 Nov 29. PMID 25432633
- [Background] Stacey FG, James EL, Chapman K, Lubans DR. Social cognitive theory mediators of physical activity in a lifestyle program for cancer survivors and carers: findings from the ENRICH randomized controlled trial. Int J Behav Nutr Phys Act. 2016 Apr 14;13:49. doi: 10.1186/s12966-016-0372-z. PMID 27075417
- [Background] Sterner RC, Sterner RM. CAR-T cell therapy: current limitations and potential strategies. Blood Cancer J. 2021 Apr 6;11(4):69. doi: 10.1038/s41408-021-00459-7. PMID 33824268
- [Background] Stout NL, Santa Mina D, Lyons KD, Robb K, Silver JK. A systematic review of rehabilitation and exercise recommendations in oncology guidelines. CA Cancer J Clin. 2021 Mar;71(2):149-175. doi: 10.3322/caac.21639. Epub 2020 Oct 27. PMID 33107982
- [Background] Suleman A, Vijenthira A, Berlin A, Prica A, Rodin D. The Use of Virtual Care in Patients with Hematologic Malignancies: A Scoping Review. Curr Oncol. 2022 Feb 7;29(2):892-900. doi: 10.3390/curroncol29020076. PMID 35200575
- [Background] Sweet SN, Michalovic E, Latimer-Cheung AE, Fortier M, Noreau L, Zelaya W, Martin Ginis KA. Spinal Cord Injury Peer Mentorship: Applying Self-Determination Theory to Explain Quality of Life and Participation. Arch Phys Med Rehabil. 2018 Mar;99(3):468-476.e12. doi: 10.1016/j.apmr.2017.08.487. Epub 2017 Sep 22. PMID 28947164
- [Background] Tallantyre EC, Evans NA, Parry-Jones J, Morgan MPG, Jones CH, Ingram W. Neurological updates: neurological complications of CAR-T therapy. J Neurol. 2021 Apr;268(4):1544-1554. doi: 10.1007/s00415-020-10237-3. Epub 2020 Nov 2. PMID 33140239
- [Background] Taylor S, Bellhouse S, Allsop M, Radford J, Yorke J. The Role of e-Health in the Delivery of Care for Patients with Hematological Cancers: A Systematic Literature Review. Telemed J E Health. 2020 Sep;26(9):1093-1105. doi: 10.1089/tmj.2019.0231. Epub 2020 Mar 24. PMID 32208067
- [Background] Thomas J, Harden A. Methods for the thematic synthesis of qualitative research in systematic reviews. BMC Med Res Methodol. 2008 Jul 10;8:45. doi: 10.1186/1471-2288-8-45. PMID 18616818
- [Background] Thompson-Leduc P, Clayman ML, Turcotte S, Legare F. Shared decision-making behaviours in health professionals: a systematic review of studies based on the Theory of Planned Behaviour. Health Expect. 2015 Oct;18(5):754-74. doi: 10.1111/hex.12176. Epub 2014 Feb 16. PMID 24528502
- [Background] Tong A, Sainsbury P, Craig J. Consolidated criteria for reporting qualitative research (COREQ): a 32-item checklist for interviews and focus groups. Int J Qual Health Care. 2007 Dec;19(6):349-57. doi: 10.1093/intqhc/mzm042. Epub 2007 Sep 14. PMID 17872937
- [Background] Tsai T, Finkelstein J. Design and Implementation of a Low-Cost Virtual Biking System Using IoT Interface. 2023 IEEE 9th World Forum on Internet of Things (WF-IoT), Aveiro, Portugal, 2023, pp. 1-7, doi: 10.1109/WF-IoT58464.2023.10539434.
- [Background] Tsai T, Finkelstein J. Using IoT Architecture for Remotely-Controlled Physical Telerehabilitation in Virtual Reality. 2024 IEEE 6th Eurasia Conference on Biomedical Engineering, Healthcare and Sustainability (ECBIOS 2024). June 14-16, 2024, Taiwan.
- [Background] Tseng YF, Wang KL, Lin CY, Lin YT, Pan HC, Chang CJ. Predictors of smoking cessation in Taiwan: using the theory of planned behavior. Psychol Health Med. 2018 Mar;23(3):270-276. doi: 10.1080/13548506.2017.1378820. Epub 2017 Sep 20. PMID 28931309
- [Background] Trinh L, Plotnikoff RC, Rhodes RE, North S, Courneya KS. Correlates of physical activity in a population-based sample of kidney cancer survivors: an application of the theory of planned behavior. Int J Behav Nutr Phys Act. 2012 Aug 6;9:96. doi: 10.1186/1479-5868-9-96. PMID 22866956
- [Background] Trinh L, Plotnikoff RC, Rhodes RE, North S, Courneya KS. Feasibility and preliminary efficacy of adding behavioral counseling to supervised physical activity in kidney cancer survivors: a randomized controlled trial. Cancer Nurs. 2014 Sep-Oct;37(5):E8-22. doi: 10.1097/NCC.0b013e3182a40fb6. PMID 24232192
- [Background] Trinh L, Plotnikoff RC, Rhodes RE, North S, Courneya KS. Changes in motivational outcomes following a supervised physical activity program with behavioral counseling in kidney cancer survivors: a pilot study. Psychooncology. 2015 Sep;24(9):1204-7. doi: 10.1002/pon.3754. Epub 2015 Jan 27. No abstract available. PMID 25628184
- [Background] Van Blarigan EL, Kenfield SA, Tantum L, Cadmus-Bertram LA, Carroll PR, Chan JM. The Fitbit One Physical Activity Tracker in Men With Prostate Cancer: Validation Study. JMIR Cancer. 2017 Apr 18;3(1):e5. doi: 10.2196/cancer.6935. PMID 28420602
- [Background] van Haren IE, Timmerman H, Potting CM, Blijlevens NM, Staal JB, Nijhuis-van der Sanden MW. Physical exercise for patients undergoing hematopoietic stem cell transplantation: systematic review and meta-analyses of randomized controlled trials. Phys Ther. 2013 Apr;93(4):514-28. doi: 10.2522/ptj.20120181. Epub 2012 Dec 6. PMID 23224217
- [Background] van Vugt M, de Wit M, Cleijne WH, Snoek FJ. Use of behavioral change techniques in web-based self-management programs for type 2 diabetes patients: systematic review. J Med Internet Res. 2013 Dec 13;15(12):e279. doi: 10.2196/jmir.2800. PMID 24334230
- [Background] Vermaete N, Wolter P, Verhoef G, Gosselink R. Physical activity, physical fitness and the effect of exercise training interventions in lymphoma patients: a systematic review. Ann Hematol. 2013 Aug;92(8):1007-21. doi: 10.1007/s00277-013-1689-1. Epub 2013 Feb 14. PMID 23408096
- [Background] Villumsen BR, Jorgensen MG, Frystyk J, Hordam B, Borre M. Home-based 'exergaming' was safe and significantly improved 6-min walking distance in patients with prostate cancer: a single-blinded randomised controlled trial. BJU Int. 2019 Oct;124(4):600-608. doi: 10.1111/bju.14782. Epub 2019 May 14. PMID 31012238
- [Background] Wei C, Finkelstein J. Comparison of Alexa Voice and Audio Video Interfaces for Home-Based Physical Telerehabilitation. AMIA Jt Summits Transl Sci Proc. 2022 May 23;2022:496-503. eCollection 2022. PMID 35854718
- [Background] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093
- [Background] Wilson HK, Wieler C, Bell DL, Bhattarai AP, Castillo-Hernandez IM, Williams ER, Evans EM, Berg AC. Implementation of the Diabetes Prevention Program in Georgia Cooperative Extension According to RE-AIM and the Consolidated Framework for Implementation Research. Prev Sci. 2024 Apr;25(Suppl 1):34-45. doi: 10.1007/s11121-023-01518-0. Epub 2023 Mar 17. PMID 36930404
- [Background] Wood J, Wallin M, Finkelstein J. Can a low-cost webcam be used for a remote neurological exam? Stud Health Technol Inform. 2013;190:30-2. PMID 23823365
- [Background] Ziegler A. Generalized Estimating Equations. Springer, 2011. ISBN 978-1-4614-0498-9.
- [Background] Zweben A, Fucito LM, O'Malley SS. Effective Strategies for Maintaining Research Participation in Clinical Trials. Drug Inf J. 2009 Jul;43(4):10.1177/009286150904300411. doi: 10.1177/009286150904300411. PMID 24311825